CLINICAL TRIAL: NCT04651231
Title: Values of Releasable Sutures in Punch Trabeculectomy Prospective Randomized Study
Brief Title: Punch Trabeculectomy Versus Classic Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, khaled hamdi elbaklish, assistant professor- ophthalmic department- faculty of medicine-Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWA000017585-FMASU R23/2017
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Eighty Patients inclusive, randomly distributed for tight flap technique group (forty patients-group A) and for loose flap technique (securing sutures) group (forty patients-group B).
Who Masked: Participant
Masking Description: The participants were masked during study time through permuted variable block randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tight flap technique group (forty patients-group A) (Active Comparator): in this arm forty patients did tight flap technique for punch trabeculectomy. At 12 o'clock 10/0 nylon monofilament stitch was used to close the apex of triangular scleral flap tightly and two releasable stitches were used at the sides of triangular scleral flap.
  Interventions: Procedure: releasable sutures in punch trabeculectomy
- loose flap technique (securing sutures) group (forty patients-group B). (Experimental): in this arm forty patients did loose flap technique for punch trabeculectomy. At 12 o'clock 10/0 nylon monofilament stitch was used to secure the edges of the flap at the apex of and two-four releasable stitches were used at the sides of triangular scleral flap in group B.
  Interventions: Procedure: releasable sutures in punch trabeculectomy

INTERVENTIONS:
Procedure: releasable sutures in punch trabeculectomy — punch trabeculectomy,scleral flap suturing
  Other Names: loose flap technique versus tight flap technique in punch trabeculectomy

SUMMARY:
Bleb failure is reduced with Punch trabeculectomy procedure. Wide sclerostomy during surgery is wanted but controllable. This can be done with single securing suture, releasable sutures and topical intraoperative mitomycin-c. Average IOP without fluctuation (risk factor) can protect the optic nerve.

DETAILED DESCRIPTION:
This is a prospective randomized study. Patients had uncontrolled glaucoma on maximum tolerated medical therapy including acetazolamide tablets were enrolled in this clinical trial and were randomized to tight flap technique group (group A) and loose flap technique group(group B). Randomization assigned 40 patients to group A and 40 patients to do group B. A total of 80 patients were enrolled in the Study between 2012 and 2014.

During trabeculectomy, Trabecular meshwork and scleral lamellae were excised made an opening with the kelly scleral punch 1.0 mm 3-5 bites. At 12 o'clock 10/0 nylon monofilament stitch was used to close the apex of triangular scleral flap tightly and two releasable stitches were used at the sides of triangular scleral flap in group A. Fig-1 At 12 o'clock 10/0 nylon monofilament stitch was used to secure the edges of the flap at the apex of and two-four releasable stitches were used at the sides of triangular scleral flap in group B. The intraocular pressure and bleb morphology were followed for one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary open-angle glaucoma
* Clinical diagnosis of pigmentary glaucoma
* Clinical diagnosis of Pseudophakic glaucoma

Exclusion Criteria:

* high risk factors for failed trabeculectomy must be present e.g. previous failed trabeculectomy surgery and active intraocular infection/ inflammation.
* Clinical diagnosis of aphakic glaucoma was excluded.
* Clinical diagnosis of glaucoma with previous ocular incisional surgery (except for clear cornea cataract surgery) were excluded.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2014-06-28 (Actual); Study Completion 2014-10-16 (Actual)

PRIMARY OUTCOMES:
postoperative intraocular pressure (IOP) | one-year follow up
  measuring IOP at first day ,first month, three months, six months, nine months,and one year after surgery frequent interval in both groups with applanation method( Goldmann applanation tonometer

SECONDARY OUTCOMES:
bleb morphology after surgery | one-year follow up
  examination of bleb formed after surgery with Silt Lamp.we comment on the bleb features on each patient in study groups as grade-1 (high elevated bleb), grade-2 (low elevated bleb), grade-3-(encysted bleb), grade-4 (flat bleb).

IPD SHARING:
Plan to Share IPD: No
Given the data in determining evidence-based medicine and evidence-based public health policies, sharing this type of data is seen as particularly important.